CLINICAL TRIAL: NCT06219252
Title: Intraoperative Aberrometry vs Conventional Introcular Lens Calculation ( Barrett Universal II / Barrett True K ), Refractive and Visual Outcomes, a Prospective Study.
Brief Title: Intraoperative Aberrometry vs Conventional Intraocular Lens Calculation, a Prospective Study.
Acronym: ORAVSCTRL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CI-005-2023
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Intraocular Lens Implantation; Cataract; Humans; Ocular, Refraction
Keywords: biometry; aberrometry; prospective study
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Masking Description: None of the patients will be informed in what group they are assigned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- ORA group (Experimental): the intraocular lens calculation in this group will be optimized by the intraoperative aberrometer (ORA)
  Interventions: Device: Intraoperative aberrometer
- Control group (Active Comparator): Barrett universal II will be used in the control group.
  Interventions: Other: Preoperative intraocular lens calculation

INTERVENTIONS:
Device: Intraoperative aberrometer — the patient intraocular lens will be optimized during the aphakic period after cataract extraction and before intraocular lens implantation, this will produce a possible change in the dioptric power of the intraocular lens
  Other Names: ORA
  Arms: ORA group
Other: Preoperative intraocular lens calculation — the intraocular lens in this group will be calculated preoperatively with Barrett Universal II formula
  Other Names: Barrett Universal II
  Arms: Control group

SUMMARY:
the goal of this intervention study is to compare prospectively the accuracy of the power calculation between both groups, the intraoperative aberrometry (ORA) vs barrett universal II preoperative calculation (control group) .

Researchers will compare ORA group vs control to see changes in spherical equivalent and uncorrected distance visual acuity

DETAILED DESCRIPTION:
Studies have described a small difference between ORA (intraoperative aberrometer) and preoperative calculation with latest generation formulas ( Barrett Universal II ), the investigators intend to compare both groups prospectively, during the process randomization and blinding of the participants will be made.

The investigators will report spherical equivalent and uncorrected distance visual acuity values at 90 days of the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* patients with senile cataract, patients undergoing phacoemulsification, complete biometric profile, axial length calculated by interferometer.

Exclusion Criteria:

* glaucoma, uncontrolled diabetic retinopathy, pseudoexfoliation syndrome, aged macular degeneration , dry eye syndrome, other ocular pathologies.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
spherical equivalent | 90 days of the postoperative period
  Spherical equivalent values at 90 days of the postoperative period

SECONDARY OUTCOMES:
uncorrected distance visual acuity | 90 days of the postoperative period
  uncorrected distance visual acuity at 90 days of the postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: ANGEL NAVA - CASTAÑEDA, MD, Principal Investigator — INSTITUTO DE OFTALMOLOGIA CONDE DE VALENCIANA
Locations (1):
- Instituto de oftalmología Fundación Conde de Valenciana, Mexico City, Cuauhtemoc, Mexico